CLINICAL TRIAL: NCT02705885
Title: Evaluation of IgY Antibody Effectiveness in Supportive Therapy of Periodontitis Patients
Brief Title: IgY Efficacy on Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Immunology Research Institute in Gifu (Industry)
Collaborators: National Hospital of Odonto-Stomatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RHM 14
Record Dates: First submitted 2015-11-25; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Periodontitis
Keywords: IgY; Periodontitis; Porphyromonas gingivalis; gingipains; Efficacy
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gingipain IgY (Experimental): Participants consume lozenges containing IgY against gingipains of Porphyromonas gingivalis
  Interventions: Dietary Supplement: lozenges containing IgY
- Placebo IgY (Placebo Comparator): Participants consume lozenges containing placebo IgY
  Interventions: Dietary Supplement: Placebo IgY

INTERVENTIONS:
Dietary Supplement: lozenges containing IgY — Patients consumed food supplement lozenges containing IgY after nonsurgical periodontal therapy
  Arms: Gingipain IgY
Dietary Supplement: Placebo IgY — Placebo IgY
  Arms: Placebo IgY

SUMMARY:
Patients visiting National Hospital of Odonto-Stomatology for treating periodontitis used a food supplement (lozenge) containing chicken egg antibody (IgY) against Porphyromonas gingivalis gingipains as an adjunct to conventional scaling and root planing (SRP). After 8 weeks the patients were examined against. Parameters including probing depth (PD), bleeding on probing (BOP), number of P. gingivalis in periodontal pockets were evaluated and compared to the control group that had used placebo lozenges.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with chronic periodontitis
* had at least 2 interproximal site with pocket depth between 3 mm to 5 mm
* nonsmokers with at least 20 natural teeth
* bone loss and bleeding on probing
* had not undergone periodontal treatments within 6 weeks before the study

Exclusion Criteria:

* patients received medication such as antibiotics or anti-inflammatory drugs within the previous 3 months
* had allergy to egg proteins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effect of anti-gingipain IgY on probing pocket depth of subjects with chronic periodontitis | 8 weeks
  Outcome measurement is probing pocket depth (PD)
Effect of anti-gingipain IgY on bleeding on probing of subjects with chronic periodontitis | 8 weeks
  Outcome measurement is bleeding on probing (BOP)

SECONDARY OUTCOMES:
Effect of anti-gingipain IgY on Porphyromonas gingivalis level of subjects with chronic periodontitis | 8 weeks
  Outcome measurement is P. gingivalis level in periodontal pockets

CONTACTS AND LOCATIONS:
Overall Officials: Thi Hong Minh Nguyen, Ph. D, Principal Investigator — National Hospital of Odonto-Stomatology